CLINICAL TRIAL: NCT07050901
Title: The Effect of Nursing Care Based on Kolcaba's Comfort Theory on the Quality of Life and Psychological Well-Being Levels of the Aged People
Brief Title: Theory of Kolcaba on the Quality of Life and Psychological Well-Being Levels of the Aged People
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Merve OZKAN (Other)
Responsible Party: Sponsor-Investigator, Merve OZKAN, PhD, Aydin Adnan Menderes University
Organization: Aydin Adnan Menderes University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Interventional studies
Record Dates: First submitted 2025-06-04; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Elderly (People Aged 65 or More); Quality of Life; Psychological Well-being; Nurse
Keywords: quailty of life; nursing; psychological well-being; elderly
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment group (Experimental): The experimental group will receive training on Nursing Care Based on Kolcaba's Comfort Theory. For the individuals in the experimental group, follow-up measurements will be made in the 1st month and 3rd month after the completion of Kolcaba's Nursing Care Based on Comfort Theory training.
  Interventions: Other: Nursing Care Based on Kolcaba's Comfort Theory
- Control group (No Intervention): The control group continued to receive the routine care

INTERVENTIONS:
Other: Nursing Care Based on Kolcaba's Comfort Theory — Kolcaba's Nursing Care Applications Based on Comfort Theory were carried out individually; each application was planned for one and a half hours, one day a week and for 8 weeks, and each session was carried out for each individual through home visits. The topics of Nursing Care Based on Kolcaba's Comfort Theory were; Physical Care Practices (2 weeks), Psychospiritual Care Practices (2 weeks), Environmental Care Practices (2 weeks) and Sociocultural Care Practices (2 weeks).
  Arms: Experiment group

SUMMARY:
A randomised controlled study will be conducted to determine the effect of nursing care based on Kolcaba's comfort theory on the quality of life and psychological well-being levels of the elderly.

DETAILED DESCRIPTION:
The aim of this study was to determine the effect of nursing care based on Kolcaba's comfort theory on the quality of life and psychological well-being levels of the elderly. This study is a randomized controlled experimental research. The population of the study consisted of 775 individuals aged 65 and over residing in Çeştepe and Tepecik neighborhoods of Efeler district of Aydın province, and the sample consisted of a total of 112 individuals, 56 in the experimental group and 56 in the control group. The data of the study were collected with the questionnaire form prepared by the researcher, Quality of Life Scale in the Elderly and Psychological Well-Being Scale in the Elderly. Each intervention was planned for one and a half hours, 1 day a week for 8 weeks, and each session was carried out individually for the experimental group through home visits. Follow-up measurements were made at the 1st month and 3rd month after the interventions of the experimental group were completed. The control group did not receive any intervention until the end of the study and follow-up measurements were performed at the 1st month and 3rd month after the first measurement. Descriptive statistical analyses, Mann Whitney U, Likelihood Ratio, Pearson chi-square and Friedman tests were used for comparisons outside normal distribution. The Kolmogorov-Smirnov test was used to evaluate normal distribution as a baseline analysis; values at p<0.05 level were considered statistically significant. Ethics committee, mukhtar's office, scale use permissions and participant written consents were obtained. When the sociodemographic characteristics of the elderly in the experimental and control groups were compared, it was found that there was a significant difference in terms of social security and having a chronic disease, in the comparison of the mean scores of the total and sub-dimensions of the Quality of Life in the Elderly Scale of the 1st and 2nd Measurement before and after the training of the elderly in the experimental and control groups; no difference was found before the training, and the mean scores of the elderly in the experimental group were higher than the control group. measurement autonomy sub-dimension, post-training 1st measurement pleasure sub-dimension, post-training 1st measurement self-actualization sub-dimension and post-training 1st measurement Quality of Life in the Elderly Scale total mean scores were higher than the control group.

When the pre-training, post-training (1st and 2nd measurements) mean scores of the Quality of Life Scale for the Elderly (total and sub-dimensions) were compared within the experimental group, a statistically significant difference was found in the self-realization sub-dimension. Furthermore, when the total mean scores of the Psychological Well-Being Scale for the Elderly were compared at the same time points within the experimental group, a statistically significant difference was observed (p < 0.05).

In the control group, when the pre-training, post-training (1st and 2nd measurements) mean scores of the Quality of Life Scale for the Elderly (total and sub-dimensions) were compared, statistically significant differences were observed in the total score, as well as in the control, autonomy, pleasure, and self-realization sub-dimensions. Additionally, a significant difference was found in the total mean scores of the Psychological Well-Being Scale for the Elderly across the same time points in the control group (p < 0.05).

In the experimental group, statistically significant increases were observed in the total score of the Quality of Life Scale and in the sub-dimensions of autonomy, pleasure, and self-realization, as well as in the scores of the Psychological Well-Being Scale following the training. Although some significant differences were also identified in certain sub-dimensions over time within the control group, the increases observed in the experimental group were more pronounced and statistically significant. These findings suggest that the training provided had a positive impact on the quality of life and psychological well-being levels of elderly individuals.

ELIGIBILITY:
Inclusion Criteria:

* Volunteered to participate in the research,
* Residing in Aydın,
* No mental disability,
* 65 years of age or older,
* At least primary school graduate (since the scales should be filled in by self-report method),
* individuals who can speak and write Turkish language were included.

Exclusion Criteria:

* individuals staying in nursing homes/nursing homes were excluded from the scope of the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
experimental group measurement | September 2023
  measurement of quality of life and psychological well-being levels of the elderly up to 5 months with a questionnaire form

SECONDARY OUTCOMES:
control group measurement | December 2023
  up to 3 months measurement of quality of life and psychological well-being levels of the elderly with a questionnaire form

CONTACTS AND LOCATIONS:
Locations (1):
- AydınAdnan Menderes University institute of health sciences, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request
Supporting Information: CSR
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.